CLINICAL TRIAL: NCT03830047
Title: Effect of nd Yag Laser in Treatment of Vulval Warts
Brief Title: Effect of Laser in Treatment of Vulval Warts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: laser
Record Dates: First submitted 2019-02-02; First posted 2019-02-05 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Vulval Wart
MeSH Terms: interventions — Lasers, Solid-State; Lasers

STUDY DESIGN:
Intervention Model Description: applying laser for treatment of vulval warts
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nd yag laser (Active Comparator): Applying nd yag laser to vulva
  Interventions: Device: nd yag laser
- Co2 laser (Sham Comparator): Applying CO2 laser to vulva
  Interventions: Device: nd yag laser

INTERVENTIONS:
Device: nd yag laser — nd yag laser will be applied on the vulval warts
  Other Names: laser beam

SUMMARY:
Vulval warts is a magor problem that affects women .

DETAILED DESCRIPTION:
The causative organism for vulval warts is human papilloma virus There are many treatment modalities that can trat these warts

ELIGIBILITY:
Inclusion Criteria:

* women who have vulval warts
* Age between 18- 40 years

Exclusion Criteria:

* warts that were previously treated by surgery or cryotherapy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females who have vulval warts
Enrollment: 40 (Estimated)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-10-15 (Estimated); Study Completion 2019-11-20 (Estimated)

PRIMARY OUTCOMES:
The number of women who will be completely cured by laser beam | within 2 months
  how laser will cure the warts

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (3):
- Egypt (3):
  - Algazeerah and Kasralainy hospital, Giza
  - Algazeerah, Giza
  - Aljazeera( Al Gazeera) hospital, Giza